CLINICAL TRIAL: NCT01515501
Title: Endoscopic Mucosal Resection for the Diagnosis of a-Ganglionosis, a Controlled Prospective Trial (EDGE Trial)
Acronym: EDGE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Branden Kuo, Instructor in Medicine, Harvard Medical School, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MGH2007p001577
Record Dates: First submitted 2012-01-11; First posted 2012-01-24 (Estimated); Last update posted 2018-08-16 (Actual); Status verified 2018-08

CONDITIONS: Constipation; Hirschsprung Disease
Keywords: Constipation; Hirschsprung Disease
MeSH Terms: conditions — Constipation; Hirschsprung Disease | interventions — Endoscopic Mucosal Resection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Endoscopic mucosal resection (Other): At time of rectal section biopsy all subjects will under go the additional intervention of an endoscopic muscosal resection.
  Interventions: Procedure: Endoscopic mucosal resection (EMR)

INTERVENTIONS:
Procedure: Endoscopic mucosal resection (EMR) — EMR uses an endoscope to take a tissue sample from the rectum. It is the same type of instrument used in a routine colonoscopy. It is hoped that this procedure will help diagnose Hirschsprung's Disease more often than by recal suction biopsy alone, which can often be unclear and result in more invasive surgery for diagnosis.

SUMMARY:
Patients undergoing routine rectal suction biopsy will undergo as part of the study an additional Endoscopic mucosal resection. The biopsy results will also be correlated with patient's clinical data including clinical history, Bristol stool scale, anorectal manometry results, and SITZ marker studies. Cost and recovery time will be compared.

DETAILED DESCRIPTION:
Background: Adult and pediatric patients presenting with chronic constipation and/or motility disorders may be referred for rectal biopsy to rule out aganglionosis or Hirschsprung's disease. The traditional diagnostic test, rectal suction biopsy, is a blind technique and is insensitive in confirming the diagnosis. Frequently, patients require subsequent referral for a surgical full thickness biopsy.

Hypothesis: Endoscopic mucosal resection (EMR) will improve the diagnostic yield for aganglionosis and decrease the need for subsequent surgical full thickness biopsy.

Methods: This is a prospective, single center, controlled investigation of EMR for the diagnosis of colonic aganglionosis / Hirschsprung's disease. Patients who are offered rectal suction biopsy will be offered enrollment. Enrolled patients will have one additional procedure (EMR) at the time of their rectal suction biopsy. Specimens will be analyzed pathologically for size, submucosal tissue adequacy, the presence of ganglionic tissue, and positivity by acetylcholinesterase staining. The adequacy of the tissue specimen, the proportion of diagnostic specimens, and the proportion of patients that would have required subsequent referral for full thickness biopsy, will be compared. Variable such as cost and recovery time will be compared. Biopsy results will be compared with patient's pre-endoscopy clinical data including their history of constipation, results of SITZ marker studies, Bristol stool scale, and anorectal manometry.

Results: The primary outcome variable will be the proportion of patients with a diagnostic specimen in each group. Secondary outcome variables will include the size of the specimen, the presence of ganglionic tissue, the presence of submucosal tissue, and the positivity of the acetylcholinesterase stain. The biopsy results will also be correlated with patient's clinical data including clinical history, Bristol stool scale, anorectal manometry results, and SITZ marker studies. Cost and recovery time will be compared.

Discussion: The proposed investigation may demonstrate that a simple endoscopic test, which uses direct visualization, can improve the diagnostic yield of rectal biopsies for Hirschsprung's disease, and spare patients an additional surgical full thickness rectal biopsy.

ELIGIBILITY:
Inclusion Criteria:

* 10 years of age or older
* offered Rectal Suction biopsy

Exclusion Criteria:

* any contraindication to general anesthesia or conscious sedation
* contraindication to endoscopy
* untreated or unmanageable coagulopathy
* thrombocytopenia (<50)
* inability to provide informed consent.

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2007-10 (Actual); Primary Completion 2012-02 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
The number of EMR Biopsies that are diagnostic specimens | One Year
  The adequacy of the tissue specimen, the proportion of diagnostic specimens, and the proportion of patients that would have required subsequent referral for full thickness biopsy, will be compared. Variable such as cost and recovery time will be compared. Biopsy results will be compared with patient's pre-endoscopy clinical data including their history of constipation, results of SITZ marker studies, Bristol stool scale, and anorectal manometry.

CONTACTS AND LOCATIONS:
Overall Officials: Braden Kuo, M.D., Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Croffie JM, Davis MM, Faught PR, Corkins MR, Gupta SK, Pfefferkorn MD, Molleston JP, Fitzgerald JF. At what age is a suction rectal biopsy less likely to provide adequate tissue for identification of ganglion cells? J Pediatr Gastroenterol Nutr. 2007 Feb;44(2):198-202. doi: 10.1097/01.mpg.0000252188.12793.ee. PMID 17255831
- [Background] Hurlstone DP, Cross SS, Drew K, Adam I, Shorthouse AJ, Brown S, Sanders DS, Lobo AJ. An evaluation of colorectal endoscopic mucosal resection using high-magnification chromoscopic colonoscopy: a prospective study of 1000 colonoscopies. Endoscopy. 2004 Jun;36(6):491-8. doi: 10.1055/s-2004-814397. PMID 15202044
- [Background] Hirose R, Hirata Y, Yamada T, Kawana T, Taguchi T, Suita S. The simple technique of rectal mucosal biopsy for the diagnosis of Hirschsprung's disease. J Pediatr Surg. 1993 Jul;28(7):942-4. doi: 10.1016/0022-3468(93)90703-n. PMID 7693906
- [Background] Pini-Prato A, Martucciello G, Jasonni V. Rectal suction biopsy in the diagnosis of intestinal dysganglionoses: 5-year experience with Solo-RBT in 389 patients. J Pediatr Surg. 2006 Jun;41(6):1043-8. doi: 10.1016/j.jpedsurg.2006.01.070. PMID 16769331